CLINICAL TRIAL: NCT02650908
Title: Does the Avivement of Suturing Area is Essential for Healing a Meniscus Lesion ?
Brief Title: Is Abrasion of the Suture Area Essential for Healing of a Meniscus Lesion?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6295
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-01

CONDITIONS: Meniscus Lesion
Keywords: Lesion; Meniscus; Avivement; Suturing area

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The most common technique involves a suture meniscus avivement with a rasp or a motorized cutter the suture zone before actual implementation of the suture. But the imperative nature of this avivement is based only on theoretical considerations. The team has an old experience in conducting meniscus sutures without avivement. It therefore seems interesting to compare results with those of literature

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients who underwent meniscal suturing with or without avivement

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent meniscal suturing with or without avivement
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Healing meniscus suturing area | For the duration of hospital stay, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France